CLINICAL TRIAL: NCT00701961
Title: The Pharmacokinetic of the Fixed-dose Combination of Mefloquine-Artesunate in Plasmodium Falciparum Malaria Infection in Pregnant Women
Brief Title: Pharmacokinetic of Mefloquine-Artesunate in Plasmodium Falciparum Malaria Infection in Pregnancy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Centre Muraz (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Prof. Umberto D'Alessandro, Parasitology Department, Institute Tropical Medicine, Antwerp, Belgium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITMP0208
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Mefloquine-artesunate; Malaria; Pregnancy; Pharmacokinetics; Sub-Saharan Africa; P falciparum malaria infection in pregnancy
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pregnat women receiving MQ-AS fixed dose combination comprised of 100 mg of artesunate and 220mg of mefloquine per tablet, dosed once daily such that mefloquine dose is approximately 8mg/kg/day for 3 days.
  Interventions: Drug: Mefloquine-artesunate
- 2 (Active Comparator): Non-pregnant women receiving MQ-AS fixed dose combination comprised of 100 mg of artesunate and 220mg of mefloquine per tablet, dosed once daily such that mefloquine dose is approximately 8mg/kg/day for 3 days.
  Interventions: Drug: Mefloquine-artesunate

INTERVENTIONS:
Drug: Mefloquine-artesunate — Mefloquine-artesunate fixed dose combination comprised of 100 mg of artesunate and 220mg of mefloquine per tablet, developed by DNDi and manufactured by farmanguinhos (Brazil).
  Other Names: MQ-AS

SUMMARY:
Malaria in pregnancy is a major public health problem in Sub-Saharan Africa. Over the past decades, P. falciparum has shown increasing resistance to chloroquine and Sulphadoxine-Pyrimethamine, which has prompted a change in treatment approach; artemisinin containing combination therapies (ACTs) are now the standard treatment of P. falciparum malaria in areas with established resistance to traditional therapies. However, a standard approach for using ACT in pregnancy does not exist in Africa, where some countries keep on using quinine, while others allow the use of ACTs. Thus, there is need of establishing the safety and efficacy of ACTs in malaria-infected pregnant women. Since the pharmacokinetic of antimalarials may be altered during pregnancy and since available pharmacokinetic data are still somewhat limited, we propose to carry out a study confirming or disproving existing pharmacokinetic data (collected in South-East Asia), before starting any larger African efficacy and safety trials. The fixed-dose combination mefloquine-artesunate (MQ-AS), developed by the Drugs for Neglected Diseases Initiative, will be used in the study, which will compare the pharmacokinetics of MQ-AS for treatment of P.falciparum in 24 pregnant women in the second and third trimesters, to the pharmacokinetics of this regimen in 24 matched non-pregnant P.falciparum infected women. The study will be carried out in Burkina Faso.

DETAILED DESCRIPTION:
Malaria during pregnancy constitutes a major public health problem in Sub-Saharan Africa, where it increases the risk of low birth weight (<2500g), infant mortality, infant morbidity during the first year of life, prematurity and infant anemia. Over the past decades, P. falciparum has shown increasing resistance to standard antimalarial therapy (chloroquine CQ and Sulphadoxine-Pyrimethamine). The inexorable development and spread of P. falciparum resistance to antimalarials has prompted a change in treatment approach; artemisinin containing combination therapies (ACTs) are now the standard treatment of P. falciparum malaria in areas with established resistance to the traditional therapies. The use of combinations reduces the theoretical likelihood of selecting resistant mutants; it is hoped that this strategy will delay the development of new resistances.

A standard approach for using ACT in pregnancy does not exist in Africa. Even if the World Health Organization endorses the use of ACTs for treatment of uncomplicated malaria in 2nd and 3rd trimesters of pregnancy, some countries keep on using quinine, while others allow the use of ACTs. These different approaches point out to the necessity of establishing the safety and efficacy of ACTs in malaria-infected pregnant women. Nevertheless, considering that the pharmacokinetic of antimalarials may be altered during pregnancy (potentially leading to under-dosing) and that the available safety and pharmacokinetic data are still somewhat limited, it is important to carry out a preliminary pharmacokinetic study confirming or disproving available data (collected in South-East Asia), before starting any larger African efficacy and safety trials.

The ACT regimen mefloquine-artesunate (MQ-AS) has recently been developed as a fixed-dose combination by the Drugs for Neglected Diseases Initiative (DNDi) and has been registered in Brazil (the country of manufacture) in 2008. Artesunate is an artemisinin derivative with a rapidly increasing positive experience in pregnancy, while Mefloquine (Lariam®) has been used for many years for both prevention and treatment of malaria, and has been shown to be safe in pregnant women. The convenient dosing afforded by a fixed drug combination makes MQ-AS a very promising candidate for use in treating pregnant women in Africa, as rescue treatment alternative to quinine. Since preliminary data suggest that the peak concentration of mefloquine is lowered in pregnant women, further studies on safety, efficacy, and dose optimization are imperative, prior to wide-spread adoption of this medicine.

Therefore, we propose to compare the pharmacokinetics of the fixed combination of MQ-AS for treatment of P.falciparum in 24 pregnant women in the second and third trimesters to the pharmacokinetics of this regimen in 24 matched non-pregnant P.falciparum infected women, in an African setting. This will allow for dose optimization in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Plasmodium falciparum monoinfection (any density)
2. At least 18 years old;
3. Haemoglobin at leats 7 g/dL;
4. Residence within the health facility catchment's area;
5. Willing to adhere to the study requirements
6. Willing to deliver in health facility
7. Ability to provide written informed consent
8. EITHER pregnant women in the 2nd or 3rd trimester (cases)or non-pregnant women between the ages of 18 and 49 years (controls).

Exclusion Criteria:

1. Pregnancy 1st trimester
2. History of known pregnancy complications or bad obstetric history such as repeated stillbirths or eclampsia;
3. Known major illnesses likely to influence pregnancy outcome including diabetes mellitus, severe renal or heart disease, or active tuberculosis;
4. Current cotrimoxazole prophylaxis or ARV treatment;
5. Any significant presenting illness that requires hospitalization, including severe malaria;
6. Intent to move out of the study catchment area before delivery or deliver at relative's home out of the catchment area.
7. Prior enrollment in the study or concurrent enrollment in another study.
8. Unable to take oral medication
9. Clear evidence of treatment with antimicrobials with antimalarial activity (erythromycin or other macrolides, co-trimoxazole or other sulfonamides, any tetracycline including doxycycline, quinolones and clindamycin) or exposure to antimalarial drugs within the week prior enrollment.
10. History of allergy or hypersensivity to interventional drugs
11. Patients taking drugs with possible interaction with study drugs (i.e. digoxin or warfarin)
12. History or family history of epilepsy or psychiatric disorder
13. Presence of signs and symptoms of severe malaria
14. Inability to tolerate oral medication (repeated vomiting, impairment of consciousness). Vomiting of any of the treatment doses will lead to exclusion from the pharmacokinetic sampling.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To estimate the pharmacokinetic of MQ-AS for treatment of P. falciparum or mixed infection in pregnant compared to non-pregnant women. | 6 months

SECONDARY OUTCOMES:
The proportion of women in each treatment group with parasitological cure at 63 days, corrected by PCR for re-infection. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tinto Halidou, PhD, Principal Investigator — Centre Muraz; Umberto D'Alessandro, MD, Study Chair — ITM Belgium
Locations (1):
- Centre Muraz, Nanoro, Burkina Faso

REFERENCES:
- [Derived] Birgersson S, Valea I, Tinto H, Traore-Coulibaly M, Toe LC, Hoglund RM, Van Geertruyden JP, Ward SA, D'Alessandro U, Abelo A, Tarning J. Population pharmacokinetics of artesunate and dihydroartemisinin in pregnant and non-pregnant women with uncomplicated Plasmodium falciparum malaria in Burkina Faso: an open label trial. Wellcome Open Res. 2019 Mar 7;4:45. doi: 10.12688/wellcomeopenres.14849.2. eCollection 2019. PMID 32025570
- [Derived] Valea I, Tinto H, Traore-Coulibaly M, Toe LC, Lindegardh N, Tarning J, Van Geertruyden JP, D'Alessandro U, Davies GR, Ward SA. Pharmacokinetics of co-formulated mefloquine and artesunate in pregnant and non-pregnant women with uncomplicated Plasmodium falciparum infection in Burkina Faso. J Antimicrob Chemother. 2014 Sep;69(9):2499-507. doi: 10.1093/jac/dku154. Epub 2014 Jun 2. PMID 24891429